CLINICAL TRIAL: NCT02560545
Title: Cannabinoids Effects on the Pain Modulation System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Head of R&D department, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: TASMC-15-LD-0001-15-CTIL
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cannabis oil (Active Comparator): Cannabis oil, 20% THC 0.2 mg/kg
  Interventions: Drug: Cannabis oil
- Placebo (Placebo Comparator): Oil
  Interventions: Drug: Cannabis oil

INTERVENTIONS:
Drug: Cannabis oil — Cannabis oil 20% THC

SUMMARY:
Effective treatment of acute pain, chronic and persistent is the most important concern in the world today. Although a variety of pain medications including anti-inflammatory painkillers and opiouids, patients continue to suffer from pain constantly. For over a century ,International committees studied the issue of cannabis, and almost uniformly recommended the use of cannabis for various medical applications ,especially those that include pain treatment.

Despite the widespread use of THC in clinical practice, there are few studies on the efficacy of THC In a double-blind, randomized trial. In addition, few studies examined the effect of THC on the experience pain in healthy subjects and most of them did not find an effect on pain experimental induced by capsain. so checking other models of pain such as thermal pain and mechanical pain in addition to checking the influence on the regulation of pain will contribute to understanding the mechanism of action of THC. Understanding the mechanism of action of THC in relieving pain will lead to predicting who will benefit from this treatment and direct patients for selection of appropriate medication according to the damaged mechanism.

ELIGIBILITY:
Inclusion Criteria:

A. Men aged 25-65. B. Were not treated with formulation contains Cannabis C. Can sign an informed consent form. D. Patients have a medical history that supports severe neuropathic pain over Three months And do not respond to other painkillers or suffer from side effects resulting from the use them E. At least moderate pain (more than 40 on a scale of 0-100 visual analogue scale). F. Did not receive epidural injection or invasive treatment in The last month before the entry to study . G. Not drinking alcohol or consuming high concentrations of opioid and Benzodiazifinim over 24 Hours before the experiment (equivalent to 40 mg morphine).

Exclusion Criteria:

A. Patients that found with serious level of anxiety in Patient Health Questionnaire (PHQ-9) . (These patients will be recommended by a doctor appointment with a psychiatrist). B.Patients with psychiatric problems or a family history of psychiatric disorders.

C.Patients with known cardiovascular problems D.Patients with neurological problems from a central source E.Patients taking blood pressure medication F.Patients who are unable to understand and follow the instruction of the study.

G.Diffuse pain syndromes from uncertain origin (like fibromyalgia) H.Alcoholism or chronic use of drugs. I.Malignant

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
evaluation of pain | 1 months
  The evaluation will be made by Questionnaire

SECONDARY OUTCOMES:
Testing of the pain and pain-modulation system | 1 months
  The testing will be made and analyzed by TSA Neurosensory Analyzer
Functional brain correlates | 1 month
  will be examined using fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- Pain Institute, Tel Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weizman L, Sharon H, Dayan L, Espaniol J, Brill S, Nahman-Averbuch H, Hendler T, Jacob G. Oral Delta-9-Tetrahydrocannabinol (THC) Increases Parasympathetic Activity and Supraspinal Conditioned Pain Modulation in Chronic Neuropathic Pain Male Patients: A Crossover, Double-Blind, Placebo-Controlled Trial. CNS Drugs. 2024 May;38(5):375-385. doi: 10.1007/s40263-024-01085-0. Epub 2024 Apr 10. PMID 38597988